CLINICAL TRIAL: NCT03605199
Title: An Open-label, Multi-center, Phase 2 Study of Denosumab in Subjects With Giant Cell Rich Tumors of Bone
Brief Title: Denosumab in Subjects With Giant Cell Rich Tumors of Bone
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, HansGelderblom, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20159990
Record Dates: First submitted 2018-06-15; First posted 2018-07-30 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Aneurysmal Bone Cysts; Giant Cell Granuloma; Osteoblastoma; Chondroblastoma; Chondromyxoid Fibroma
Keywords: denosumab; giant cell rich tumor of bone
MeSH Terms: conditions — Bone Cysts, Aneurysmal; Granuloma, Giant Cell; Osteoblastoma; Chondroblastoma | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Denosumab active treatment (Experimental): Denosumab active treatment
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab will be given in a dose of 120mg subcutaneously (SC) on day 1 of every 4 week cycle with a loading dose of 120mg SC on days 8 and 15 of the first cycle.
  Other Names: Xgeva

SUMMARY:
An open-label, multi-center, phase 2 study of the efficacy of denosumab in subjects with giant cell rich tumors of bone. The population will consist of subjects with the following tumor types: aneurysmal bone cysts (ABC), giant cell granuloma (GCG) and other giant cell rich lesions (primary bone, non-malignant).

DETAILED DESCRIPTION:
In this phase 2 single arm trial subjects with giant cell rich tumors that would require morbid surgery OR with tumors that have recurred after previous surgery will be treated with denosumab. The primary objectives of the study are to evaluate avoidance of surgery and performance of less morbid surgical procedure compared with the planned surgical procedure at baseline in subjects with salvageable giant cell rich tumors during the study. For subjects with unsalvageable tumors the objective is to evaluate disease control (radiological response assessed by combined RECIST, PET, inverse Choi when available and/or no progression at 1 year (based on disease assessment) in combination with stable pain score defined as ≤ 1 point increase on 'worst pain' question in BPI-SF).

Surgical resection may occur at any time during the study based on the clinical judgement of the Investigator. For subjects that undergo surgical tumor resection, denosumab treatment will be discontinued after surgery. In all other cases, denosumab treatment continues for a maximum of up to 3 years, or until confirmation of disease progression, the Investigator's or Sponsor's recommendation of discontinuation, the subject's decision to discontinue for any reason or administration of any of the prohibited therapies listed in the study protocol. For subjects that continue to show clinical benefit after 3 years of treatment with denosumab, ongoing treatment outside of study protocol is optional after discussion with Amgen.

For assessment of histopathological response and for translational research purposes a tumor sample will be requested either during study or at the EOT (surgical sample only for the subject group that has undergone surgery).

During the time the study is still open, re-treatment may be allowed for subjects who demonstrated a response to denosumab and are currently not receiving denosumab treatment (e.g., in the case of recurrent disease while subject is in the safety follow-up phase or subjects that have completed the study and have later experienced disease progression). The re-treatment decision including the use of the loading dose and discontinuation of therapy will be handled on a case-by-case basis; prior authorization from the Sponsor is required. Subjects must meet all inclusion/exclusion criteria prior to being considered for re-treatment, with the exception of the exclusion criterium of previous denosumab treatment. The same subject number will be assigned to avoid bias.

Overall in total approximately 60 subjects with giant cell rich tumors that would require morbid surgery or with tumors that have recurred after previous surgery will be included. The investigators expect 50% of subjects will have salvageable giant cell rich tumors and the remaining 50% of subjects to have unsalvageable giant cell rich tumors.

The population will consist of subjects with the following cohorts according to tumor type:

* Aneurysmal bone cysts (ABC), ~ approximately 40 subjects
* Giant Cell Granuloma (GCG) and other giant cell rich lesions (primary bone, non-malignant), ~ approximately 20 subjects

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven giant cell rich tumor:

  * Aneurysmal bone cysts (ABC)
  * Giant cell granuloma (GCG)
  * Other giant cell rich lesions (primary bone, non-malignant, pathology and radiology to be reviewed during multidisciplinary meeting LUMC)
* Patients with surgically unsalvageable disease (e.g., sacral, spinal giant cell rich tumors, or multiple lesions including pulmonary metastases) OR patients whose planned surgery includes joint resection, limb amputation, hemipelvectomy or surgical procedure resulting in severe morbidity
* Measurable evidence of active disease within 1 year before study enrollment
* Albumin-adjusted serum calcium level ≥ 2.0 mmol/L (8.0 mg/dL)
* Aged 18 years and up and skeletally mature
* ECOG performance status 0, 1 or 2
* Written signed informed consent

Exclusion Criteria:

* Known or suspected current diagnosis of classic GCTB
* Known or suspected current diagnosis of underlying malignancy including but not limited to high-grade sarcoma, osteosarcoma, fibrosarcoma, malignant giant cell sarcoma
* Known or suspected current diagnosis of brown cell tumor of hyperparathyroidism, Paget's disease or cherubism
* Known or suspected current diagnosis of primary soft tissue tumor with invasion of the bone
* Known diagnosis of other malignancy within the past 5 years (patients with definitively treated basal cell carcinoma and cervical carcinoma in situ are permitted)
* Previous treatment with denosumab (with the exception of patients eligible for re-treatment with denosumab after completing this study)
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction
* Non-healed dental/oral surgery
* Planned invasive dental procedure for the course of the study
* Known hypersensitivity to denosumab
* Known hypersensitivity to products to be administered during the study (calcium and/or vitamin D)
* Currently receiving other specific treatment for giant cell rich tumors of bone (e.g., radiation, chemotherapy or embolization)
* Concurrent bisphosphonate treatment
* Major surgery less than 4 weeks prior to start of treatment
* Treatment with other investigational device or drug 30 days prior to study enrollment
* Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before enrollment
* Patient is pregnant or breast feeding, or planning to become pregnant within 5 months after the EOT visit
* Female patient of child bearing potential is not willing to use a highly effective method of contraception during treatment and for 5 months after the EOT visit
* Patient has any kind of disorder that compromises the ability of the patient to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy (proportion of subjects who do not require surgery during the study) | Continuous monitoring until surgery of max treatment duration of 3 years.
  (For subgroup of subjects with salvageable tumors):The proportion of subjects who do not require surgery during the study.
Efficacy (proportion of subjects undergoing the planned versus performed type of surgery during the study) | Continuous monitoring until surgery of max treatment duration of 3 years.
  (For subgroup of subjects with salvageable tumors): The proportion of subjects undergoing the planned versus performed type of surgery during the study.
Efficacy (Radiological response) | Imaging to be performed every 3 months. Up to maximum duration of treatment of 3 years.
  (For subgroup of subjects with UNsalvageable tumors) Combined endpoint: 1. Disease control:
  o Radiological response assessed by combined RECIST, PET, inverse Choi criteria when available
Efficacy (disease progression based on clinical disease assessment) | Clinical disease assessment performed every 4 weeks. Up to maximum duration of treatment of 3 years.
  (For subgroup of subjects with UNsalvageable tumors) Combined endpoint: 2. Disease control:
  o No progression at 1 year (based on clinical disease assessment)
Efficacy (combined pain scores) | Questionnaires on pain to be performed every 4 weeks. Up to maximum duration of treatment of 3 years.
  (For subgroup of subjects with UNsalvageable tumors) Combined endpoint: 3. Stable pain score, defined as ≤ 1 point increase on 'worst pain' question in Brief Pain Inventory - Short Form (BPI-SF, measures pain severity on a scale of 0 to 10 [10 being worse pain], and pain interference on a scale of 0 to 10 [10 being complete interference], scores are averaged in total test score).

SECONDARY OUTCOMES:
Toxicity according to CTCAE v 4.03 | Assessed every 4 weeks up to 3 years.
  - Frequency of adverse events (AEs), as determined by Common Terminology Criteria for Adverse Events (CTCAE) v. 4.03 criteria
Disease recurrence after denosumab followed by surgery. | Follow-up every 6-12 months after end of treatment, up to 5 years max.
  The proportion of subjects with disease recurrence after denosumab followed by surgery during the study.
Symptomatic improvement. | Questionnaires to be performed every 4 weeks during first 6 months on treatment, after 6 months assessment is every 12 weeks. Up to 3 years.
  Symptomatic improvement in the Brief Pain Inventory - Short Form (BPI-SF, measures pain severity on a scale of 0 to 10 [10 being worse pain], and pain interference on a scale of 0 to 10 [10 being complete interference], scores are averaged in total test score).
Symptomatic improvement. | Questionnaires to be performed every 4 weeks during first 6 months on treatment, after 6 months assessment is every 12 weeks. Up to 3 years.
  Symptomatic improvement in the European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire C30 (EORTC QLC-30, 28 questions regarding interference of disease with QoL ranging from 1 'not at all' to 4 'very much', 2 questions regarding QoL raging from 1 'very poor' to 7 'excellent', scores are averaged in total test score)
Time to surgery | Continuous monitoring, clinical assessment every 4 weeks during treatment and every 6-12 months after end of treatment up to max of 5 years.
  Time in months
Time to recurrence after surgery (for patients with salvageable disease) | Continuous monitoring, clinical assessment every 4 weeks during treatment and every 6-12 months after end of treatment up to max of 5 years
  Time in months
Progression free survival | Continuous monitoring, clinical assessment every 4 weeks during treatment and every 6-12 months after end of treatment up to max of 5 years
  Time in months
Overall survival. | Continuous monitoring, clinical assessment every 4 weeks during treatment and every 6-12 months after end of treatment up to max of 5 years
  Time in months

OTHER OUTCOMES:
Translational research. | Pathology samples once during study or at end of treatment (surgery), max duration of 3 years.
  Translational research on tumor material, including proportion of subjects with pathological response for subjects undergoing surgery.

CONTACTS AND LOCATIONS:
Overall Officials: AJ Gelderblom, Prof, Principal Investigator — Leiden University Medical Center
Locations (3):
- Centre Léon Bérard, Lyon, France
- Istituto Ortopedico Rizzoli, Bologna, Italy
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lipplaa A, Schreuder WH, Pichardo SEC, Gelderblom H. Denosumab in Giant Cell Rich Tumors of Bone: An Open-Label Multicenter Phase II Study. Oncologist. 2023 Nov 2;28(11):1005-e1104. doi: 10.1093/oncolo/oyad196. PMID 37449658